CLINICAL TRIAL: NCT00000868
Title: A Phase I Safety and Immunogenicity Trial of Orally Administered Live Attenuated Recombinant Salmonella Typhi CVD 908 Delta-asd (pW57-asd+) Expressing HIV-1 LAI gp120 (VVG 203) and Parenterally Administered HIV-1 MN rgp120 in Alum in HIV-1-Uninfected Volunteers
Brief Title: A Study to Evaluate the Safety and Effectiveness of HIV-1 LAI gp120 (an HIV Vaccine) Given With or Without HIV-1 MN rgp120 (Another HIV Vaccine) to HIV-Negative Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 028; 10578 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Vaccines, Synthetic; HIV-1; Administration, Oral; AIDS Vaccines; HIV Seronegativity; HIV Envelope Protein gp120; Recombination, Genetic; Salmonella typhi; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — Aluminum Hydroxide; MF59 oil emulsion

INTERVENTIONS:
Biological: Salmonella typhi CVD 908-HIV-1 LAI gp 120 (VVG 203)
Biological: Aluminum hydroxide
Biological: MF59
Biological: rgp120/HIV-1MN

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of giving healthy volunteers a new oral HIV vaccine which has been incorporated into a bacterial cell. This oral vaccine (HIV-1 LAI gp120) will be given with or without a different injected HIV vaccine (HIV-1 MN rgp120).

Vaccines are preparations that are introduced into the body to try to prevent infection or create resistance to infection. This study examines a new oral vaccine to see if it can improve the immune system's ability to fight the HIV virus when given alone or with another injected vaccine.

DETAILED DESCRIPTION:
Although recent advances have been made in antiviral therapy for AIDS, there is no cure for HIV-1 infection or AIDS, and drug therapy is too expensive for most affected populations. The development of safe, effective vaccines to prevent HIV-1 infection and AIDS worldwide is a global priority. One promising approach in the development of HIV-1 vaccines utilizes live vaccines as vectors to express HIV-1 antigens. The potential advantages of the live vector approach include the ability of live vector recombinants to induce long-lasting humoral and cell-mediated immunity (particularly neutralizing antibody and CD8+ cytotoxic T-cell activity) and the relatively low cost of production. Moreover, live vector recombinant vaccines administered orally might be able to stimulate the production of secretory IgA vaccine-specific antibodies locally at relevant mucosal sites.

Part I of this study is conducted as an open-label, dose-escalation trial. The first 5 volunteers (Group A) receive a single oral dose of Salmonella typhi CVD 908-HIV-1 LAI gp 120 (VVG203). If no typhoid fever-like illness is seen in these volunteers during at least 14 days of follow-up, the next 5 patients (Group B) receive a single dose of VVG203. If this higher dose is well-tolerated, Phase II of the study is initiated once all Phase I volunteers have been assessed for safety for at least 21 days. [AS PER AMENDMENT 11/07/97: Groups A and B are expanded to 10 patients each.] Part II of this study is a randomized, placebo-controlled, double-blind trial. Nine volunteers are randomized to each of treatment groups, with oral VVG203 given alone or sequentially with HIV-1 SF-2 rgp 120 in MF59 (SF) given intramuscularly. [AS PER AMENDMENT 11/07/97: Randomization is to VVG 203 alone or sequentially with HIV-1 MN rgp120 in alum (MN).] A total of 3 vaccinations are administered within each 9-person cohort, 1 volunteer serves as a control and receives a sodium bicarbonate buffer rather than VVG203 or a vaccine placebo rather than SF. Group C receives VVG at Month 0 and SF at Months 2 and 6. Group D receives VVG at Months 0, 2, and 6. Group E receives SF at Months 0 and 2 and VVG at Month 6. [AS PER AMENDMENT 11/07/97: MN is given in place of SF in all Groups C, D, and E.]

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 18-50 years old.
* Are HIV-negative.
* Are healthy and have a normal history and physical exam.
* Agree to practice abstinence or use of effective birth control for 1 month before and during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of immune deficiency, chronic illness, or autoimmune disease.
* Have received immunosuppressive medications, blood products, trial drugs, immunoglobulins, or an HIV or typhoid vaccine.
* Have a history of severe allergic reactions.
* Have had prior suicidal attempts or have a psychiatric condition or job commitments which would prevent you from completing the study.
* Have a history of cancer (unless the cancer has been successfully cured), gallbladder disease, typhoid fever, migraines or other severe headaches, cardiac valve defects, or congenital heart disease.
* Have active syphilis or tuberculosis.
* Are allergic to certain medications.
* Are pregnant or breast-feeding.
* Have household contact with infants or persons who are pregnant, immunodeficient, or HIV-positive.
* Are unavailable for 12 months of follow-up.
* Have hepatitis B.
* Have a history of injection drug use within 12 months of enrollment or have higher or intermediate risk sexual behavior.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27
Dates: Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Clements, Study Chair; D Schwartz, Study Chair
Locations (1):
- JHU AVEG, Baltimore, Maryland, United States